CLINICAL TRIAL: NCT01636024
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single and Multiple Ascending Inhaled Doses of AZD7594 in Healthy Male Volunteers
Brief Title: To Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ascending Doses of Inhaled AZD7594
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D3740C00001
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Safety; Pharmacokinetics; Pharmacodynamics of AZD7594
Keywords: Phase 1,; healthy volunteers,; safety,; tolerability,; pharmacokinetics,; pharmacodynamics,; single ascending dose study,; multiple
MeSH Terms: interventions — velsecorat

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Subjects will participate in 1 of up to 9 groups in Part A (single ascending dose part) or 1 of 4 groups in Part B (multiple ascending dose part). Ratio of subjects receiving AZD7594 versus placebo is 6:2 in part A and 6:3 in Part B.
  Interventions: Drug: AZD7594
- 2 (Placebo Comparator): Subjects will participate in 1 of up to 9 groups in Part A or 1 of 4 groups in Part B. Ratio of subjects receiving AZD7594 versus placebo is 6:2 in part A and 6:3 in Part B.
  Interventions: Drug: Placebo to match

INTERVENTIONS:
Drug: AZD7594 — Suspension inhaled via Spira nebuliser
  Arms: 1
Drug: Placebo to match — Matching placebo inhaled via Spira nebuliser
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety profile and look at levels of AZD7594 and biomarkers in blood when the drug is administered inhaled to healthy subjects

DETAILED DESCRIPTION:
A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single and Multiple Ascending Inhaled Doses of AZD7594 in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18-45 years inclusive with suitable veins for cannulation or repeated vein puncture
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weight between 50 and 100 kg (inclusive)
* Be able to inhale from the Spira nebuliser used in the study
* Be willing to use a condom with spermicide to prevent pregnancy and drug exposure of a female partner

Exclusion Criteria:

* History of any clinically significant disease or disorder
* Current smokers
* Any clinically relevant abnormal findings

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety profile in terms of adverse events, ECG, blood pressure, pulse, physical examination, body temperature, haematology, clinical chemistry, urinalysis and spirometry. | Screening to 13 days post last dose.
  No statistical tests will be performed

SECONDARY OUTCOMES:
Single dose pharmacokinetics (PK) of AZD7594 in terms of : Cmax, tmax, λz, t1/2λz, AUC(0-last), AUC(0-24), AUC, CL/F, Vz/F, MRT, Cmax/D, AUC/D, AUC(0-24)/D. | pre-dose and at 5, 15 and 30 minutes and 1, 2, 4, 6, 9, 12, 18, 24, 36 and 48 hours post-dose. From cohort four 72 and 96 hours post-dose samples will also be taken.
  Cmax- max plasma concentration;tmax-Time to max plasma concentration,λz- terminal rate constant;t1/2λz - Terminal half-life;AUC(0-24) - Area under the plasma concentration time curve from zero to 24 hours;AUC- Area under the plasma concentration
Multiple dose PK of AZD7594 in terms of: Cmax, tmax, λz, t1λz, AUC(0-last), AUC(0-24), AUC, CL/F, Vz/F, MRT, Cmax/D, AUC/D,AUC(0-24)/D, Cavg, %Fluctuation, Rac(Cmax) and Rac(AUC(0-24) and time-dependency (AUC(0-24) and AUC) | pre-dose and at 5, 15 and 30 min and 1, 2, 4, 6, 9, 12, 18, 24, 48, 72 hours and 96 h post-dose. Days 6-15: Pre-dose samples only.From day 16: pre-dose and 5, 15 and 30 min and 1, 2, 4, 6, 9, 12, 18, 24, 36 and 48 h post-dose.
  CL/F- Apparent plasma clearance;Vz/F- Apparent volume of distribution during terminal phase; MRT- Mean residence time; Rac Cmax-Accumulation ratio of Cmax
Pharmacodynamics of AZD7594 following a single dose in terms of: 24-hour plasma cortisol | screening and on the dosing day at the following time points 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24. On the dosing day also at 36 and 48 hours post dose.
Pharmacodynamics of AZD7594 following a multiple doses in terms of: 24-hour plasma cortisol | screening and days 1 and 16 at the following time points 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 and 24 hours. On day 1 also at 36 and 48 hours.
Pharmacodynamics of AZD7594 following multiple doses in terms of: Plasma cortisol after adrenocorticotropic hormone stimulation | screening and day 17 at 30 minutes and 1 hour post tetracosactide injection
Pharmacodynamics of AZD7594 following multiple doses in terms of: Plasma dehydroepiandrosterone sulphate, plasma 4β-OH-cholesterol, and plasma osteocalcin | screening and day 17

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, MD, Study Director — AstraZeneca R&D, Molndal Sweden
Locations (1):
- Research Site, London, UK, United Kingdom